CLINICAL TRIAL: NCT05207254
Title: Research on the Application of Artificial Intelligence Ultrasonic Recognition
Brief Title: Research on the Application of Artificial Intelligence Ultrasonic Recognition Technology in Difficult Airway Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2021-T356-2
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2021-12

CONDITIONS: Difficult Airways

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult airway: C-L≥3 grade
  Interventions: Diagnostic Test: Ultrasonic test
- none difficult airway: C-L<3 grade
  Interventions: Diagnostic Test: Ultrasonic test

INTERVENTIONS:
Diagnostic Test: Ultrasonic test — Ultrasonic test to the patient's head, neck and jaw area.

SUMMARY:
Although there is no related research on the evaluation of difficult airways by ultrasound features based on artificial intelligence, the investigators guess that the evaluation of ultrasound features based on artificial intelligence can make further breakthroughs in difficult airway early warning systems. Therefore, this project intends to use AI technology to extract and analyze the ultrasound features of the subjects, evaluate the correlation between the ultrasound features of the subjects and the occurrence of difficult airways, and construct possible diagnostic models to evaluate AI ultrasound feature recognition in the prediction of difficult airways. The effect and application value of this method are expected to be more intelligent and accurate for early warning of difficult airways in clinical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification is 1-3
* Patients who intend to undergo tracheal intubation under general anesthesia
* Age ≥ 18 years old

Exclusion Criteria:

* Patients with speech communication and cooperation barriers;
* Patients with open head and neck trauma
* Patients with cervical spine fractures or cervical spine diseases;
* Emergency surgery;
* Patients who are allergic to related drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults who intend to undergo tracheal intubation under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosed as a difficult airway | 0-10minutes after intubation
  Cormack-Lehane was used for grading the best glottic view. In grade the entire glottis was visible; in grade 2 a portion of the glottis was visible; in grade 3 only the epiglottis could be seen; and in grade 4 the epiglottis was not visible. A score of 3-4 indicated difficult video laryngoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 9Th Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No